CLINICAL TRIAL: NCT02260141
Title: Treating Alzheimer's and Dementia With D-ribose
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to get adequate enrollment
Sponsor: Practitioners Alliance Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN- ALZ001
Record Dates: First submitted 2014-10-05; First posted 2014-10-09 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2017-10

CONDITIONS: Alzheimers; Dementia
MeSH Terms: conditions — Dementia | interventions — Ribose

STUDY DESIGN:
Intervention Model Description: Single arm pilot study using ribose for alzheimers
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with d-ribose (Experimental): Treatment with ribose 5 gm TID
  Interventions: Dietary Supplement: d-ribose

INTERVENTIONS:
Dietary Supplement: d-ribose — giving ribose in those with a diagnosis of Alzheimer's and/or dementia

SUMMARY:
To study the effectiveness of d-ribose in treating Alzheimer's and Dementia

DETAILED DESCRIPTION:
Clinical experience and the pathophysiology of Alzheimer's, including neuronal insulin resistance, suggests that ribose improves clinical outcomes. This study will add ribose 5 gm 3 X day for 8 weeks to monitor outcomes in a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Alzheimer's and/or dementia with a Mini Mental Status Exam ( MMSE) score over 12 or being ambulatory and able to travel outside the home with assistance.
* Must have a caregiver living with them.

Exclusion Criteria:

* Overt and severe causes of secondary dementia such as metastatic brain cancers, or severe overt infectious encephalopathies or severe autoimmune illness.
* Also, severe life threatening illnesses which would make them unlikely to be alive after 6-12 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
ADAS-ADL | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- PAN, Kailua, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No